CLINICAL TRIAL: NCT02203747
Title: Patient Perception of Visual Distortions
Status: Completed | Type: Observational
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Other Study IDs: TIOL-201-VPAS
Record Dates: First submitted 2014-07-10; First posted 2014-07-30 (Estimated); Results first posted 2015-12-22 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-09

CONDITIONS: Cataract; Astigmatism
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pseudophakic implanted with toric IOL: Subjects bilaterally implanted with toric IOL
  Interventions: Other: Administration of patient self-assessment
- Pseudophakic implanted with non-toric IOL: Subjects bilaterally implanted with non-toric IOL
  Interventions: Other: Administration of patient self-assessment

INTERVENTIONS:
Other: Administration of patient self-assessment

SUMMARY:
The purpose of this study is to evaluate visual distortions reported by pseudophakic patients.

ELIGIBILITY:
Inclusion Criteria:

* Corneal astigmatism of at least 0.75 diopters
* Bilaterally-implanted with monofocal toric intraocular lenses in both eyes or with monofocal non-toric intraocular lenses in both eyes
* At least one month postoperative from second-eye surgery
* Ability to understand, read and write English to give consent and complete study questionnaire
* Availability, willingness, and sufficient cognitive awareness to comply with examination procedures and study visits
* Sign informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Any ocular pathology of clinical significance, as determined by the investigator, other than regular corneal astigmatism, that may affect visual outcomes or influence subjective ocular visual symptoms
* Patient is pregnant or is lactating
* Participation in any other clinical trial during the last 30 days prior to study enrollment or concurrent participation in any other ongoing clinical trial
* Other protocol-defined exclusion criteria may apply

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Bilaterally-implanted pseudophakic subjects over 22 years of age with astigmatism who meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact AMO for Trial Locations, Santa Ana, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pseudophakic Implanted With Toric IOL: Subjects implanted with bilateral toric IOL
  Administration of patient self-assessment
- Pseudophakic Implanted With Non-toric IOL: Subjects implanted with bilateral non-toric IOL
  Administration of patient self-assessment
Period: Overall Study
Arm/Group | Pseudophakic Implanted With Toric IOL | Pseudophakic Implanted With Non-toric IOL
Started | 45 | 34
Completed | 45 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pseudophakic Implanted With Toric IOL | Pseudophakic Implanted With Non-toric IOL | Total
Number analyzed (Participants) | 45 | 34 | 79
Age, Categorical [Number; unit: participants] — Total participants in the "Pseudophakic implanted with toric IOL" group is 45, but age was not reported for one subject.
  participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 8 | 9 | 17
    >=65 years | 36 | 25 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.39 (8.34) | 69.68 (11.08) | 70.64 (9.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 18 | 41
  Male | 22 | 16 | 38
Region of Enrollment [Number; unit: participants]
  United States | 45 | 34 | 79

OUTCOME MEASURES:

1. Primary Outcome: Visual Distortion Symptoms
Description: Subjective rating of visual distortion symptoms under overall conditions at baseline. Rating scale consisted of the following categories: "did not experience" (rating = 0), "mild" (rating = 1), "moderate" (rating = 2), or "severe" (rating = 3), therefore, the lower values represent the best outcome. The minimum score was 0 and the maximum score was 3.
Time Frame: Baseline
Population: Of the 45 subjects in the "Pseudophakic implanted with toric IOL" group, one (#102) was excluded due to a protocol deviation (improper method used to simulate visual distortion).
Measure: Mean (Standard Deviation); unit: rating of visual distortion symptoms
Groups:
- Pseudophakic Implanted With Toric IOL: Subjects implanted with toric IOL
  Administration of patient self-assessment
- Pseudophakic Implanted With Non-toric IOL: Subjects implanted with non-toric IOL
  Administration of patient self-assessment
Arm/Group | Pseudophakic Implanted With Toric IOL | Pseudophakic Implanted With Non-toric IOL
Number analyzed (Participants) | 44 | 34
rating of visual distortion symptoms
  Lines that tilt/slant | 0.89 (1.13) | 0.38 (0.65)
  Flat surfaces appear curved | 0.64 (0.97) | 0.38 (0.55)
  objects appear further away/closer than they are | 0.66 (0.78) | 0.56 (0.70)
  Objects have different size/shape | 0.75 (0.99) | 0.62 (0.92)
  physical discomfort related to vision | 0.73 (0.90) | 0.56 (0.75)

2. Primary Outcome: Visual Distortion Symptoms
Description: as for outcome 1
Time Frame: 1 week
Population: Of the 45 subjects in the "Pseudophakic implanted with toric IOL" group, one (#307) was excluded due to a protocol deviation (subject visit was completed outside of the protocol-defined visit interval).
Measure: Mean (Standard Deviation); unit: rating of visual distortion symptoms
Arm/Group | Pseudophakic Implanted With Toric IOL | Pseudophakic Implanted With Non-toric IOL
Number analyzed (Participants) | 44 | 34
rating of visual distortion symptoms
  Lines that tilt/slant | 0.82 (0.95) | 0.65 (0.85)
  Flat surfaces appear curved | 0.64 (0.87) | 0.38 (0.6)
  objects appear further away/closer than they are | 0.64 (0.78) | 0.47 (0.61)
  Objects have different size/shape | 0.61 (0.84) | 0.47 (0.79)
  physical discomfort related to vision | 0.59 (0.92) | 0.47 (0.79)

ADVERSE EVENTS:
Arm/Group | Pseudophakic Implanted With Toric IOL | Pseudophakic Implanted With Non-toric IOL
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/34
Other Adverse Events (participants affected / at risk) | 0/45 | 2/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pseudophakic Implanted With Toric IOL (N=45) | Pseudophakic Implanted With Non-toric IOL (N=34)
Headache with dizziness and nausea (Surgical and medical procedures) | 0 (0) | 1 (1) — Subject reported feeling nausea with a headache and dizziness hours after astigmatism induction
Achiness and pressure (Immune system disorders) | 0 (0) | 1 (1) — Subject experienced achiness and eye pressure after experiencing a lupus flare-up, unrelated to study procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Trial Agreement